CLINICAL TRIAL: NCT00028899
Title: A Dose Finding Study of the Safety of Gemtuzumab Ozogamicin Combined With Conventional Chemotherapy for Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Monoclonal Antibody Plus Chemotherapy in Treating Young Patients With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: AAML00P2; COG-AAML00P2 (Other: Children's Oncology Group); CDR0000069145 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; previously treated myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Asparaginase; Cytarabine; Gemtuzumab; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: asparaginase
Drug: cytarabine
Drug: gemtuzumab ozogamicin
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as gemtuzumab ozogamicin can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with combination chemotherapy may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combining gemtuzumab ozogamicin with combination chemotherapy in treating children who have relapsed or refractory acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and maximum tolerated dose of gemtuzumab ozogamicin in combination with conventional chemotherapy in patients with relapsed or refractory acute myeloid leukemia or myelodysplastic syndromes.
* Determine the efficacy of this regimen in these patients.
* Correlate the likelihood of leukemic blast cells to undergo apoptosis in vitro with the efficacy of this regimen in these patients.
* Correlate drug resistance as manifested by dye efflux or multiple drug resistance-1 expression by leukemic blast cells with the efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study of gemtuzumab ozogamicin. Patients are assigned by cohort to 1 of 2 treatment regimens.

* Regimen A: Patients receive cytarabine IV over 2 hours every 12 hours on days 1-4, mitoxantrone IV over 1 hour on days 3-6, and gemtuzumab ozogamicin IV over 2 hours on day 7.
* Regimen B: Patients receive cytarabine IV over 3 hours every 12 hours on days 1, 2, 8, and 9, asparaginase intramuscularly on days 2 and 9, and gemtuzumab ozogamicin IV over 2 hours on day 3.

Cohorts of 3-6 patients receive de-escalating doses of gemtuzumab ozogamicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose below that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed monthly for 6 months, every 2 months for 6 months, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 52 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary acute myeloid leukemia (AML) or myelodysplastic syndromes

  * Relapsed (remission duration less than 1 year) OR
  * Failed induction (failed to achieve an initial complete response)
* Patients with AML as a second malignant neoplasm allowed provided no other prior therapy for AML
* M2 or M3 bone marrow aspirate at time of study entry
* No Fanconi's anemia
* No known CNS leukemia

PATIENT CHARACTERISTICS:

Age:

* 21 and under

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 times normal
* AST or ALT less than 2.5 times upper limit of normal
* No history of veno-occlusive disease of the liver defined as weight increase of more than 5% over baseline and serum bilirubin greater than 5 mg/dL within 20 days after receipt of chemotherapy

Renal:

* Creatinine no greater than 1.5 times normal OR
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) at least 70 mL/min OR
* Equivalent GFR by institutional normal range

Cardiovascular:

* Shortening fraction more than 27% by echocardiogram or normal for institution OR
* Ejection fraction more than 50% by MUGA

Other:

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 180 days since prior hematopoietic stem cell transplantation

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2002-07; Primary Completion 2006-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | Length of study

SECONDARY OUTCOMES:
Toxicity
  Toxicity will be monitored through study chair notification and end course reports
Remission Rate | Length of study
  The remission rate in each arm will be estimated by the proportion of patients who achieved remission among patients who received GMTZ at the MTD level.
Prognostic Factor Analysis
  The predictive value of the likelihood of leukemia blast cells to undergo apoptosis and drug resistance of leukemia blast cells will be assessed by logistic regression

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aplenc, MD, MSCE, Study Chair — Children's Hospital of Philadelphia
Locations (76):
- United States (70):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Children's Hospital of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (5):
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec

REFERENCES:
- [Result] Aplenc R, Alonzo TA, Gerbing RB, Lange BJ, Hurwitz CA, Wells RJ, Bernstein I, Buckley P, Krimmel K, Smith FO, Sievers EL, Arceci RJ; Children's Oncology Group. Safety and efficacy of gemtuzumab ozogamicin in combination with chemotherapy for pediatric acute myeloid leukemia: a report from the Children's Oncology Group. J Clin Oncol. 2008 May 10;26(14):2390-3295. doi: 10.1200/JCO.2007.13.0096. PMID 18467731